CLINICAL TRIAL: NCT07381426
Title: Efficacy and Safety of Ferric Citrate in Iron Deficiency Anemia During the Second Trimester of Pregnancy in Bangladesh: A Randomized Controlled Trial
Brief Title: Ferric Citrate in Iron Deficiency Anemia During Pregnancy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dhaka Medical College (Other)
Collaborators: Sir Salimullah Medical College and Midford Hospital (Unknown); Mugdha Medical College and Hospital (Unknown); Shaheed Suhrawardy Medical College and Hospital (Unknown)
Responsible Party: Principal Investigator, Arifa Sharmin Maya, Assistant Professor, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/291
Record Dates: First submitted 2026-01-04; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Anemia
Keywords: Anemia; Iron deficiency
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — ferric citrate; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric citrate (Experimental): Oral ferric citrate 210 mg (providing 210 mg elemental iron daily), administered once daily for 8 weeks.
  Interventions: Drug: Ferric citrate 210 mg
- Ferrous fumarate (Active Comparator): Oral Ferrous fumarate 200 mg (providing 132 mg elemental iron daily), administered twice daily for 12 weeks or until delivery, whichever occurs earlier.
  Interventions: Drug: Ferrous fumarate 200 mg

INTERVENTIONS:
Drug: Ferric citrate 210 mg — Oral ferric citrate 210 mg (providing 210 mg elemental iron daily), administered once daily for 8 weeks.
  Arms: Ferric citrate
Drug: Ferrous fumarate 200 mg — Oral Ferrous fumarate 200 mg (providing 132 mg elemental iron daily), administered twice daily for 12 weeks or until delivery, whichever occurs earlier.
  Arms: Ferrous fumarate

SUMMARY:
Maternal anemia remains a significant public health concern in low and middle income countries including Bangladesh, contributing to adverse maternal and neonatal outcomes. Despite the widespread use of oral ferrous fumarate, gastrointestinal intolerance and suboptimal adherence remain persistent challenges, indicating the need for alternative iron formulations with improved efficacy and safety profiles. Hence, this study aims to evaluate the efficacy and safety of oral ferric citrate compared to oral ferrous fumarate in the management of maternal iron deficiency anemia during second trimester of pregnancy.

This phase 3, open-label, two-arm, parallel-group randomized controlled trial will be conducted among pregnant women aged 18-35 years, with gestational age between 13 and 26 weeks, diagnosed with moderate to severe iron deficiency anemia (hemoglobin 7-9.9 g/dL and serum ferritin <30 μg/L). Exclusion criteria are non-iron deficiency anemia, multiple pregnancy, severe comorbidities, and recent intravenous iron therapy. Eligible participants will be randomized in a 1:1 ratio to receive either oral ferric citrate 210 mg (210 mg elemental iron) once daily for 8 weeks or oral ferrous fumarate 200 mg (66 mg elemental iron) twice daily for 12 weeks or until delivery, whichever occurs earlier.

The primary endpoint is the change in maternal hemoglobin concentration from baseline to week 4 of randomization. Secondary endpoints include maternal outcome such as prevalence of anemia and iron deficiency at 36 weeks gestation and at 6 weeks postpartum, changes in maternal health-related quality of life (assessed by EQ-5D-5L), incidence of severe anemia requiring transfusion, and serious maternal medical events and neonatal outcomes such as birth weight, placental weight, birth weight percentiles, rates of low birth weight, abortion, stillbirth, preterm birth, and cord blood hemoglobin and ferritin levels, as well as infant hemoglobin and iron indices at 6 weeks of age. Safety endpoints will include incidence of adverse events, serious adverse events, maternal sick visits during the follow-up period.

Ethical approval for this trial was obtained from the institutional review boards of Dhaka Medical College, and written informed consent will be secured from all participants prior to enrollment. The findings from this trial are expected to inform clinical guidelines by establishing whether ferric citrate offers a clinically advantageous alternative to Ferrous fumarate for managing iron deficiency anemia during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 to 35 years.
* Gestational age between 13 and 26 completed weeks, confirmed by last menstrual period and/or early ultrasound dating.
* Diagnosed with moderate to severe iron deficiency anemia (IDA), defined as:

Hemoglobin concentration between 7.0 g/dL and <9.9 g/dL, and Serum ferritin concentration <30 μg/L

* Singleton intrauterine pregnancy confirmed by ultrasonography.
* Willing to comply with study procedures and follow-up schedule up to 6 weeks postpartum.
* Euthyroid or euthyroid with medications
* Normal in anomaly scan
* Received ANC check up duly
* History of folic acid intake in ANC visit
* Willing to conduct delivery at the study center or at a facility within the study catchment area.
* No known plans to leave the study area before completion of follow-up.

Exclusion Criteria:

* Known hypersensitivity or intolerance to ferric citrate, ferrous fumarate, or any excipients in the formulations.
* Presence of non-iron deficiency anemia (e.g., megaloblastic anemia, hemoglobinopathies, hemolytic anemia, anemia of chronic disease) estimated by PBF
* Baseline hemoglobin concentration <7.0 g/dL or requiring urgent transfusion according to the best clinical judgement of the consultants
* Serum ferritin ≥30 μg/L at baseline.
* Severe concurrent medical conditions including:

Chronic kidney disease (Stage 3 or higher) Decompensated liver disease Active tuberculosis or other chronic infections Diagnosed malignancy

* Pre-existing preeclampsia, or eclampsia, or gestational hypertension
* Gestational diabetes or type 2 diabetes mellitus in the current pregnancy.
* Multiple pregnancy (e.g., twins, triplets).
* Gastrointestinal conditions affecting iron absorption (e.g., inflammatory bowel disease, celiac disease, previous gastric or intestinal surgery).
* Use of intravenous iron therapy within previous 2 weeks of the present trial.
* Any other condition which, in the opinion of the investigator, may jeopardize the participant's safety or interfere with study outcomes or compliance.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 680 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration | 4 weeks
  Change in maternal hemoglobin concentration (g/dL)

SECONDARY OUTCOMES:
Anemia | 36 weeks of gestation and 6 weeks postpartum
  Prevalence of maternal anemia (Hb <11g/dL)
Iron deficiency | 36 weeks of gestation and 6 weeks postpartum
  Prevalence of maternal iron deficiency (serum ferritin concentration <30 μg/L)
Health-related quality of life | 4 weeks
  Change in maternal health-related quality of life (HRQoL) will be assessed using the EuroQol five-dimension, five-level questionnaire (EQ-5D-5L), a standardized instrument that evaluates five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a five-level ordinal scale ranging from level 1 (no problems) to level 5 (extreme problems), generating a five-digit health state that represents the respondent's self-reported health status.
  Raw EQ-5D-5L health states will subsequently be converted into a single summary index score using the country-specific value set for Bangladesh. The EQ-5D-5L index score ranges from values below 0, representing health states considered worse than death, to 1.0, representing full health. Higher index scores indicate better health-related quality of life. Changes in the EQ-5D-5L index score will be used to quantify changes in maternal HRQoL over the study period.
Severe anemia | 6 weeks postpartum
  Incidence of severe anemia requiring blood transfusion during gestation, delivery, or the puerperium
Serious maternal medical events | 6 weeks postpartum
  Incidence of serious maternal medical events, including:
  Antepartum or postpartum hemorrhage Sepsis or septic shock Intensive care unit (ICU) admission Prolonged hospital stay Wound infection confirmed by positive growth in culture of wound swab Maternal mortality
Neonatal birth weight | At birth
  Neonatal birth weight will be measured at birth (in grams)
Placental weight | At birth
  Placental weight will be measured after delivery (in grams)
Gestational age-adjusted birth weight | At birth
  Gestational age-adjusted birth weight will be measured at birth (in grams)
Incidence of abortion | through study completion, an average of 20 weeks
  Incidence of abortion
Incidence of stillbirth | During delivery
  Incidence of stillbirth
Incidence of preterm birth | During delivery
  Incidence of preterm birth
Cord venous blood hemoglobin concentration | At birth
  Cord venous blood hemoglobin concentration (g/dL) will be measured from umbilical cord blood samples collected immediately after delivery
Cord venous blood ferritin concentration | At birth
  Cord venous blood ferritin concentration (ng/mL) will be measured from umbilical cord blood samples collected immediately after delivery.
Infant hemoglobin concentration | 6 weeks after birth
  Infant hemoglobin concentration (g/dL) will be measured from peripheral venous blood samples collected at the 6-week of age
Infant serum ferritin concentration | 6 weeks after birth
  Infant serum ferritin concentration (ng/mL) will be measured from peripheral venous blood samples collected at 6 weeks of age

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
IPD will be shared on a reasonable request to the PI.